CLINICAL TRIAL: NCT07122596
Title: EFFICACY OF PROLONGED INFUSION MEROPENEM IN CRITICALLY ILL PAEDIATRIC INTENSIVE CARE PATIENTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pakistan Navy Station Shifa Hospital (Other)
Responsible Party: Principal Investigator, Nadia Iqbal, POSTGRADUATE TRAINEE, Pakistan Navy Station Shifa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNS-PG -2024-001 to 2024-150
Record Dates: First submitted 2025-08-01; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Bacterial Infection
Keywords: INFECTION; SEPSIS; BACTERIA; BACTERIAL; INTENSIVE CARE; PICU; PAEDIATRIC ICU; ICU; MEROPENEM; PROLONGED INFUSION; STANDARD INFUSION; EXTENDED
MeSH Terms: conditions — Sepsis; Bacterial Infections; Infections

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to receive either prolonged infusion or standard infusion of meropenem to compare efficacy in critically ill pediatric patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged Infusion Group (PIG) (Experimental): Drug: Meropenem (Prolonged Infusion)
  Dose: As per body weight and infection severity, following standard pediatric dosing guidelines
  Frequency: Every 8 hours (three times daily)
  Route: Intravenous (IV) infusion
  Duration: 7 days
  Other Names: Meropenem prolonged infusion
  Arm Description:
  Participants receive meropenem administered as a prolonged intravenous infusion over an extended period, instead of standard infusion duration.
  Interventions: Drug: Meropenem Infusion
- Standard Infusion Group (SIG) (Active Comparator): Drug: Meropenem (Standard Infusion) Dose: As per body weight and infection severity, following standard pediatric dosing guidelines Frequency: Every 8 hours (three times daily) Route: Intravenous (IV) infusion Duration: 7 days Other Names: Meropenem standard infusion
  Arm Description:
  Participants receive meropenem administered via standard intravenous infusion duration as per usual hospital protocol.
  Interventions: Drug: Meropenem Infusion

INTERVENTIONS:
Drug: Meropenem Infusion — Inclusion Criteria:
  * 1 month to 16 years old
  * Bacterial Infection (suspected or known) Admitted to PICU with suspected or known bacterial infection
  * Prescribed intravenous meropenem
  * Informed consent obtained from parent/guardian
  Exclusion Criteria:
  * Known allergy to carbapenems
  * Severe renal impairment (eGFR < 30 mL/min/1.73 m²)
  * Use of other investigational antibiotics at the same time
  * Prematurely Terminating the Treatment or Early Discharge Against Medical Advice Age Range: 1 month to 16 years old Gender: BOTH Sample Size (Number of participants): 150

SUMMARY:
As a broad-spectrum carbapenem, meropenem is one of the most commonly used antibiotics for critically ill pediatric patients who have severe infections. The time-dependent bactericidal activity of is consistent with the possibility that this bactericidal activity can be optimized by continuous or prolonged infusion of the drug, which would keep the drug concentration above the MIC for longer. Despite the increasing use in adult critically ill patients, the use of this process is not widely utilized in pediatric ICUs (PICUs).

With the growing concern of antimicrobial resistance, especially in children, the need for well-demonstrated dosing strategies for antimicrobials has never been more critical. Extended infusions of meropenem may provide better therapeutic effects in children by using the maximum amount of drug exposure, as well as less selection of resistance. This trial was conducted to compare the efficacy of prolonged infusion of meropenem in the critically ill visiting pediatric population, aimed at generating evidence for dosing approach in PICU.

DETAILED DESCRIPTION:
. Background and Rationale As a broad-spectrum carbapenem, meropenem is one of the most commonly used antibiotics for critically ill pediatric patients who have severe infections. The time-dependent bactericidal activity of is consistent with the possibility that this bactericidal activity can be optimized by continuous or prolonged infusion of the drug, which would keep the drug concentration above the MIC for longer. Despite the increasing use in adult critically ill patients, the use of this process is not widely utilized in pediatric ICUs (PICUs).

With the growing concern of antimicrobial resistance, especially in children, the need for well-demonstrated dosing strategies for antimicrobials has never been more critical. Extended infusions of meropenem may provide better therapeutic effects in children by using the maximum amount of drug exposure, as well as less selection of resistance. This trial was conducted to compare the efficacy of prolonged infusion of meropenem in the critically ill visiting pediatric population, aimed at generating evidence for dosing approach in PICU.

Objectives

Primary Objective:

• To evaluate the efficacy of prolonged infusion meropenem in comparison to standard infusion in critically ill pediatric patients admitted to the Pediatric Intensive Care Unit (PICU).

Secondary Objectives:

* To compare the clinical success rate between prolonged infusion and standard infusion of meropenem.
* To assess the infection clearance rate in patients receiving prolonged infusion versus standard infusion of meropenem.
* To determine the time to clinical improvement in critically ill pediatric patients treated with prolonged infusion compared to standard infusion.
* To evaluate the safety and tolerability of prolonged infusion meropenem in the PICU setting.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 16 years

Admitted to the Pediatric Intensive Care Unit (PICU) with suspected or confirmed bacterial infection

Prescribed intravenous meropenem

Informed written consent obtained from parent or legal guardian

Exclusion Criteria:

* Known allergy or hypersensitivity to carbapenem antibiotics

Severe renal impairment (eGFR < 30 mL/min/1.73 m²)

Concurrent use of other investigational antibiotics

Treatment terminated early or patient discharged against medical advice

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical success rate by Day 7 | Day 1 to Day 7 of treatment
  Defined as complete resolution of infection-related signs and symptoms, normalization of laboratory values (e.g., WBC count, CRP), and clinical stability in critically ill pediatric patients receiving either prolonged or standard meropenem infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Iqbal, MBBS, FCPS PEADS, Principal Investigator — Pakistan Navy Station Shifa Hospital
Locations (1):
- Pns Shifa Hospital, Karachi., Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policies and ethical considerations regarding patient confidentiality. Access to patient-level data is restricted to the study team to ensure data privacy and compliance with local regulations.